CLINICAL TRIAL: NCT01886105
Title: Combination of External Beam Radiotherapy With 153Sm-EDTMP to Treat High Risk Osteosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and loss of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1322; NA_00075773 (Other: JHM IRB)
Record Dates: First submitted 2013-06-04; First posted 2013-06-25 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Osteosarcoma
Keywords: Osteosarcoma; Osteogenic Sarcoma; Sarcoma; Bone Cancer
MeSH Terms: conditions — Osteosarcoma; Sarcoma; Bone Neoplasms | interventions — samarium Sm-153 lexidronam; Samarium; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SmEDTMP/Autologous Stem Cell Infusion/RT (Experimental): DAY 1 Tracer dose 153Sm-EDTMP administration (1 mCi/kg) SPECT/High-resolution CT at 4 hours. SPECT/CT (low resolution) at 24 and 48 hrs
  DAY 7 Individualized treatment dose 153Sm-EDTMP administration (max 30 mCi/kg) SPECT scans at 4, 24 and 48 hours
  DAY 21 (2 weeks following treatment dose) Auto-Stem cell infusion
  DAY 40 (approx. two weeks after stem cell rescue) Initiate EBT upon count recovery
  1 MONTH following completion of all therapy Response assessment with repeat imaging (CT/MRI, Tc-99m bone scan) 18F-MISO/FDG PET
  Interventions: Drug: Sm-EDTMP; Other: Autologous Stem Cell Infusion; Radiation: External Beam Radiotherapy

INTERVENTIONS:
Drug: Sm-EDTMP — Subjects receive a "tracer" infusion of Samarium-153 EDTMP at 1 mCi/kg. 3D dosimetry using SPECT images are obtained post "tracer" infusion to determine the distribution of dose delivered to the tumor and surrounding normal tissues. "Tracer" activity will be applied to development of the external beam radiation (EBT) planning. Second "treatment" infusion of Samarium will then be implemented. Maximum activity administered will be 30 mCi/kg.
  Other Names: Samarium; 153Sm-EDTMP
Other: Autologous Stem Cell Infusion — Administered 14 days after "Treatment" infusion of Samarium-153 EDTMP.
  Other Names: Stem Cells
Radiation: External Beam Radiotherapy — The radiotherapy portion of the combined plan will be delivered according to the judgement of the treating radiation oncologist. The total dose to be used will be modified based on surrounding tissue tolerances as evidenced by Samarium infusion and SPECT image planning.
  After the "treatment" infusion, SPECT scans will again be performed to confirm the total dose delivered and subsequently adjust the EBT portion of the treatment plan, as necessary.
  Other Names: Radiation

SUMMARY:
The primary goal of this study will be to examine tumor response after radiation treatment via a combination of Samarium-153 EDTMP and external beam radiotherapy.

DETAILED DESCRIPTION:
Samarium tracer infusion of 1 mCi/kg administered. SPECT images wil be used to determine the distribution of dose delivered to the tumor. This information will be used to determine target doses of external beam radiotherapy. The treatment infusion of Samarium, 30 mCi/kg, will be administered and dosimetry will confirm total dose delivered, and information will be used to finalize doses of external beam radiotherapy. Approximately 14 days after treatment infusion, autologous stem cells infusion is administered. Radiotherapy will be delivered according to the judgement of the treating radiation oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 13 and 65 years of age, inclusive
* Must have unresectable primary tumor or metastases
* Must have measurable disease that is demonstrated by positive Tc-99m Bone Scan. Not all lesions must be positive on bone scan.
* Creatinine clearance >70ml/min/1.73m2
* ANC >500/mm3
* Platelets >50,000/mm3
* Life expectancy > 8 weeks
* Karnofsky performance status >50%
* Stem cell product collected prior to the infusion of Samarium must be available, either by peripheral stem cell mobilization or bone marrow harvest prior to trial entry.

Exclusion Criteria:

* Patient may not be pregnant or breastfeeding.
* Patients who have received prior radiotherapy to all areas of current active disease are not eligible.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2017-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ladle, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FRANCIS KC, PHILLIPS R, NICKSON JJ, WOODARD HQ, HIGINBOTHAM NL, COLEY BL. Massive preoperative irradiation in the treatment of osteogenic sarcoma in children; a preliminary report. Am J Roentgenol Radium Ther Nucl Med. 1954 Nov;72(5):813-8. No abstract available. PMID 13207496
- [Background] Jenkin RD, Allt WE, Fitzpatrick PJ. Osteosarcoma. An assessment of management with particular reference to primary irradiation and selective delayed amputation. Cancer. 1972 Aug;30(2):393-400. doi: 10.1002/1097-0142(197208)30:23.0.co;2-2. No abstract available. PMID 4506001
- [Background] Kang CH, Ferguson-Miller S, Margoliash E. Steady state kinetics and binding of eukaryotic cytochromes c with yeast cytochrome c peroxidase. J Biol Chem. 1977 Feb 10;252(3):919-26. PMID 14138
- [Background] LEE ES, MACKENZIE DH. OSTEOSARCOMA. A STUDY OF THE VALUE OF PREOPERATIVE MEGAVOLTAGE RADIOTHERAPY. Br J Surg. 1964 Apr;51:252-74. doi: 10.1002/bjs.1800510405. No abstract available. PMID 14138245
- [Background] Singh A, Holmes RA, Farhangi M, Volkert WA, Williams A, Stringham LM, Ketring AR. Human pharmacokinetics of samarium-153 EDTMP in metastatic cancer. J Nucl Med. 1989 Nov;30(11):1814-8. PMID 2478681
- [Background] Winderen M, Kjonniksen I, Fodstad O. Pronounced therapeutic effect of samarium 153-ethylenediaminetetramethylene phosphonate in an orthotopic human osteosarcoma tibial tumor model. J Natl Cancer Inst. 1995 Feb 1;87(3):221-2. doi: 10.1093/jnci/87.3.221. No abstract available. PMID 7707409
- [Background] Lattimer JC, Corwin LA Jr, Stapleton J, Volkert WA, Ehrhardt GJ, Ketring AR, Anderson SK, Simon J, Goeckeler WF. Clinical and clinicopathologic response of canine bone tumor patients to treatment with samarium-153-EDTMP. J Nucl Med. 1990 Aug;31(8):1316-25. PMID 2384798
- [Background] Milner RJ, Dormehl I, Louw WK, Croft S. Targeted radiotherapy with Sm-153-EDTMP in nine cases of canine primary bone tumours. J S Afr Vet Assoc. 1998 Mar;69(1):12-7. doi: 10.4102/jsava.v69i1.802. PMID 9646255
- [Background] Aas M, Moe L, Gamlem H, Skretting A, Ottesen N, Bruland OS. Internal radionuclide therapy of primary osteosarcoma in dogs, using 153Sm-ethylene-diamino-tetramethylene-phosphonate (EDTMP). Clin Cancer Res. 1999 Oct;5(10 Suppl):3148s-3152s. PMID 10541356
- [Background] Turner JH, Claringbold PG, Hetherington EL, Sorby P, Martindale AA. A phase I study of samarium-153 ethylenediaminetetramethylene phosphonate therapy for disseminated skeletal metastases. J Clin Oncol. 1989 Dec;7(12):1926-31. doi: 10.1200/JCO.1989.7.12.1926. PMID 2585026
- [Background] Turner JH, Claringbold PG. A phase II study of treatment of painful multifocal skeletal metastases with single and repeated dose samarium-153 ethylenediaminetetramethylene phosphonate. Eur J Cancer. 1991;27(9):1084-6. doi: 10.1016/0277-5379(91)90297-q. PMID 1720321
- [Background] Collins C, Eary JF, Donaldson G, Vernon C, Bush NE, Petersdorf S, Livingston RB, Gordon EE, Chapman CR, Appelbaum FR. Samarium-153-EDTMP in bone metastases of hormone refractory prostate carcinoma: a phase I/II trial. J Nucl Med. 1993 Nov;34(11):1839-44. PMID 8229221
- [Background] Bruland OS, Skretting A, Solheim OP, Aas M. Targeted radiotherapy of osteosarcoma using 153 Sm-EDTMP. A new promising approach. Acta Oncol. 1996;35(3):381-4. doi: 10.3109/02841869609101655. PMID 8679270
- [Background] Franzius C, Bielack S, Flege S, Eckardt J, Sciuk J, Jurgens H, Schober O. High-activity samarium-153-EDTMP therapy followed by autologous peripheral blood stem cell support in unresectable osteosarcoma. Nuklearmedizin. 2001 Dec;40(6):215-20. PMID 11797510
- [Background] Anderson PM, Wiseman GA, Dispenzieri A, Arndt CA, Hartmann LC, Smithson WA, Mullan BP, Bruland OS. High-dose samarium-153 ethylene diamine tetramethylene phosphonate: low toxicity of skeletal irradiation in patients with osteosarcoma and bone metastases. J Clin Oncol. 2002 Jan 1;20(1):189-96. doi: 10.1200/JCO.2002.20.1.189. PMID 11773169
- [Background] Loeb DM, Garrett-Mayer E, Hobbs RF, Prideaux AR, Sgouros G, Shokek O, Wharam MD Jr, Scott T, Schwartz CL. Dose-finding study of 153Sm-EDTMP in patients with poor-prognosis osteosarcoma. Cancer. 2009 Jun 1;115(11):2514-22. doi: 10.1002/cncr.24286. PMID 19338063
- [Background] Loeb DM, Hobbs RF, Okoli A, Chen AR, Cho S, Srinivasan S, Sgouros G, Shokek O, Wharam MD Jr, Scott T, Schwartz CL. Tandem dosing of samarium-153 ethylenediamine tetramethylene phosphoric acid with stem cell support for patients with high-risk osteosarcoma. Cancer. 2010 Dec 1;116(23):5470-8. doi: 10.1002/cncr.25518. Epub 2010 Aug 16. PMID 20715156
- [Background] Ciernik IF, Niemierko A, Harmon DC, Kobayashi W, Chen YL, Yock TI, Ebb DH, Choy E, Raskin KA, Liebsch N, Hornicek FJ, Delaney TF. Proton-based radiotherapy for unresectable or incompletely resected osteosarcoma. Cancer. 2011 Oct 1;117(19):4522-30. doi: 10.1002/cncr.26037. Epub 2011 Mar 29. PMID 21448934
- [Background] Yang QC, Zeng BF, Dong Y, Shi ZM, Jiang ZM, Huang J. Overexpression of hypoxia-inducible factor-1alpha in human osteosarcoma: correlation with clinicopathological parameters and survival outcome. Jpn J Clin Oncol. 2007 Feb;37(2):127-34. doi: 10.1093/jjco/hyl137. Epub 2007 Jan 19. PMID 17237146
- [Background] Padhani AR, Krohn KA, Lewis JS, Alber M. Imaging oxygenation of human tumours. Eur Radiol. 2007 Apr;17(4):861-72. doi: 10.1007/s00330-006-0431-y. Epub 2006 Oct 17. PMID 17043737
- [Background] Koh WJ, Bergman KS, Rasey JS, Peterson LM, Evans ML, Graham MM, Grierson JR, Lindsley KL, Lewellen TK, Krohn KA, et al. Evaluation of oxygenation status during fractionated radiotherapy in human nonsmall cell lung cancers using [F-18]fluoromisonidazole positron emission tomography. Int J Radiat Oncol Biol Phys. 1995 Sep 30;33(2):391-8. doi: 10.1016/0360-3016(95)00170-4. PMID 7673026
- [Background] Rajendran JG, Wilson DC, Conrad EU, Peterson LM, Bruckner JD, Rasey JS, Chin LK, Hofstrand PD, Grierson JR, Eary JF, Krohn KA. [(18)F]FMISO and [(18)F]FDG PET imaging in soft tissue sarcomas: correlation of hypoxia, metabolism and VEGF expression. Eur J Nucl Med Mol Imaging. 2003 May;30(5):695-704. doi: 10.1007/s00259-002-1096-7. Epub 2003 Mar 11. PMID 12632200
- [Background] Rajendran JG, Mankoff DA, O'Sullivan F, Peterson LM, Schwartz DL, Conrad EU, Spence AM, Muzi M, Farwell DG, Krohn KA. Hypoxia and glucose metabolism in malignant tumors: evaluation by [18F]fluoromisonidazole and [18F]fluorodeoxyglucose positron emission tomography imaging. Clin Cancer Res. 2004 Apr 1;10(7):2245-52. doi: 10.1158/1078-0432.ccr-0688-3. PMID 15073099
- [Background] Hicks RJ, Rischin D, Fisher R, Binns D, Scott AM, Peters LJ. Utility of FMISO PET in advanced head and neck cancer treated with chemoradiation incorporating a hypoxia-targeting chemotherapy agent. Eur J Nucl Med Mol Imaging. 2005 Dec;32(12):1384-91. doi: 10.1007/s00259-005-1880-2. Epub 2005 Aug 26. PMID 16133382
- [Background] Hobbs RF, McNutt T, Baechler S, He B, Esaias CE, Frey EC, Loeb DM, Wahl RL, Shokek O, Sgouros G. A treatment planning method for sequentially combining radiopharmaceutical therapy and external radiation therapy. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1256-62. doi: 10.1016/j.ijrobp.2010.08.022. Epub 2010 Oct 13. PMID 20950958
- [Background] Hobbs RF, Sgouros G. Calculation of the biological effective dose for piecewise defined dose-rate fits. Med Phys. 2009 Mar;36(3):904-7. doi: 10.1118/1.3070587. PMID 19378750

RESULTS

PARTICIPANT FLOW:
Groups:
- SmEDTMP/Autologous Stem Cell Infusion/RT: Samarium tracer infusion of 1 mCi/kg administered. SPECT images wil be used to determine the distribution of dose delivered to the tumor. This information will be used to determine target doses of external beam radiotherapy. The treatment infusion of Samarium, 30 mCi/kg, will be administered and dosimetry will confirm total dose delivered, and information will be used to finalize doses of external beam radiotherapy. Approximately 14 days after treatment infusion, autologous stem cells infusion is administered. Radiotherapy to be delivered according to the judgement of the treating radiation oncologist.
Period: Overall Study
Arm/Group | SmEDTMP/Autologous Stem Cell Infusion/RT
Started | 4
Completed | 1
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: Individual patients
Groups:
- SmEDTMP/Autologous Stem Cell Infusion/RT: Samarium tracer infusion of 1 mCi/kg administered. SPECT images wil be used to determine the distribution of dose delivered to the tumor. This information will be used to determine target doses of external beam radiotherapy. The treatment infusion of Samarium, 30 mCi/kg, will be administered and dosimetry will confirm total dose delivered, and information will be used to finalize doses of external beam radiotherapy. Approximately 14 days after treatment infusion, autologous stem cells infusion is administered. Radiotherapy will be delivered according to the judgement of the treating radiation oncologist.
Arm/Group | SmEDTMP/Autologous Stem Cell Infusion/RT
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 23 [11 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treated Participants With 6-month Progression Free Survival
Description: Percentage of patients with high-risk osteogenic sarcoma, treated with high-dose Samarium-153 EDTMP and external beam radiotherapy, without progression at 6 months.
Time Frame: 6 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SmEDTMP/Autologous Stem Cell Infusion/RT
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Short and Long-term Side Effects of Combined Infusional Samarium-153 EDTMP and External Beam Radiotherapy as Assessed by Number of Participants With Toxicity
Description: Number of patients experiencing any Grade 3-4 toxicity, as defined by CTCAE v4.0 and RTOG Cooperative Group Common Toxicity Criteria, during the trial intervention and follow-up.
Time Frame: Up to 48 months
Measure: Count of Participants; unit: Participants
Groups:
- SmEDTMP/Autologous Stem Cell Infusion/RT: Samarium tracer infusion of 1 mCi/kg administered. SPECT images wil be used to determine the distribution of dose delivered to the tumor. This information will be used to determine target doses of external beam radiotherapy. The treatment infusion of Samarium, 30 mCi/kg, will be administered and dosimetry will confirm total dose delivered, and information will be used to finalize doses of external beam radiotherapy. Approximately 14 days after treatment infusion, autologous stem cells infusion is administered. Radiotherapy will be delivered according to the judgement of the treating radiation oncologist.
  External Beam Radiotherapy: The radiotherapy portion of the combined plan will be delivered according to the judgement of the treating radiation oncologist. The total dose to be used will be modified based on surrounding tissue tolerances as evidenced by Samarium infusion and SPECT image planning.
Arm/Group | SmEDTMP/Autologous Stem Cell Infusion/RT
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: up to 4 months
Description: No patients who enrolled on the trial survived longer than 4 months. Toxicities were graded according to CTCAE v4.0 and the RTOG Cooperative Group Common Toxicity Criteria, and attributable toxicities grade 3 or higher were recorded.
Arm/Group | SmEDTMP/Autologous Stem Cell Infusion/RT
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmEDTMP/Autologous Stem Cell Infusion/RT (N=4)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Pain from tumor requiring admission for IV pain medications.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Shortness of breath and bronchitis admitting for antibiotics
Hospitalization/Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory distress from tumor compression of airways, bleeding during airway stenting procedure leading to death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmEDTMP/Autologous Stem Cell Infusion/RT (N=4)
Nausea (Gastrointestinal disorders) | 2 (2) — Nausea grade 2 or greater
Anemia (Blood and lymphatic system disorders) | 2 (3) — Grade 2 or greater
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) — Grade 2 or greater
Pain (Psychiatric disorders) | 1 (6) — Grade 2 or greater

LIMITATIONS AND CAVEATS:
The study had low enrollment - 4 patients. Those that did enroll had very late stage disease and the therapy provided on this trial was the last therapy given for all 4 patients. Of the patients that began therapy, only 1 completed planned therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT01886105/Prot_SAP_000.pdf